CLINICAL TRIAL: NCT02677896
Title: A Multinational, Phase 3, Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study of Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus ADT in Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Brief Title: A Study of Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus ADT in Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Acronym: ARCHES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9785-CL-0335; 2015-003869-28 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Hormone Sensitive Prostate Cancer
Keywords: Androgen Deprivation Therapy (ADT); Metastatic hormone sensitive prostate cancer; Xtandi; Enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Enzalutamide + Androgen Deprivation Therapy (ADT) (Experimental): Participants received 160 mg enzalutamide orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. Eligible participants who received enzalutamide during double-blind treatment period and provided informed consent to take part in open-label period continued to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or Luteinizing hormone-releasing hormone (LHRH) agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
  Interventions: Drug: Enzalutamide
- Placebo + Androgen Deprivation Therapy (ADT) (Placebo Comparator): Participants received matching placebo orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
  Interventions: Drug: Placebo
- Placebo followed by Enzalutamide (Experimental): Eligible participants who received enzalutamide matching placebo during double-blind treatment period and provided informed consent to take part in open-label period switched to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: Xtandi
  Arms: Enzalutamide + Androgen Deprivation Therapy (ADT); Placebo followed by Enzalutamide
Drug: Placebo — Oral
  Arms: Placebo + Androgen Deprivation Therapy (ADT)

SUMMARY:
The purpose of this study was to evaluate the efficacy of enzalutamide plus androgen deprivation therapy (ADT) as measured by radiographic progression-free survival (rPFS) based on central review. The study also evaluated the safety of enzalutamide plus ADT in mHSPC.

DETAILED DESCRIPTION:
Following unblinding at the end of the double-blind period and demonstration of a statistically significant advantage of enzalutamide over placebo when added to ADT as assessed by the primary endpoint of rPFS, subjects were eligible to transition to an open-label portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of signing informed consent.
* Subject is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell or small cell histology.
* Subject has metastatic prostate cancer documented by positive bone scan (for bone disease) or metastatic lesions on computed tomography (CT) or magnetic resonance imaging (MRI) scan (for soft tissue). Subjects whose disease spread is limited to regional pelvic lymph nodes are not eligible.
* Once randomized at day 1, subject must maintain ADT with an LHRH agonist or antagonist during study treatment or have a history of bilateral orchiectomy (i.e., medical or surgical castration).
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Inclusion Criteria for Open-Label Extension:

* Subject received randomized double-blind treatment in ARCHES
* Subject has not met any of the discontinuation criteria in the main ARCHES protocol
* Subject is willing to maintain ADT with LHRH agonist or antagonist or has had a bilateral orchiectomy.
* Subject is able to swallow enzalutamide capsules whole and to comply with study requirements throughout the study
* Subject and subject's female partner agree to follow contraception and sperm donation requirements in main protocol

Exclusion Criteria:

* Subject has received any prior pharmacotherapy, radiation therapy or surgery for metastatic prostate cancer (the following exceptions are permitted):

  * Up to 3 months of ADT with LHRH agonists or antagonists or orchiectomy with or without concurrent antiandrogens prior to day 1, with no radiographic evidence of disease progression or rising PSA levels prior to day 1;
  * Subject may have 1 course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 4 weeks prior to day 1;
  * Up to 6 cycles of docetaxel therapy with final treatment administration completed within 2 months of day 1 and no evidence of disease progression during or after the completion of docetaxel therapy;
  * Up to 6 months of ADT with LHRH agonists or antagonists or orchiectomy with or without concurrent antiandrogens prior to day 1 if subject was treated with docetaxel, with no radiographic evidence of disease progression or rising PSA levels prior to day 1;
  * Prior ADT given for < 39 months in duration and > 9 months before randomization as neoadjuvant/adjuvant therapy.
* Subject had a major surgery within 4 weeks prior to day 1.
* Subject received treatment with 5-α reductase inhibitors (finasteride, dutasteride) within 4 weeks prior to day 1.
* Subject received treatment with estrogens, cyprotoerone acetate or androgens within 4 weeks prior to day 1.
* Subject received treatment with systemic glucocorticoids greater than the equivalent of 10 mg per day of prednisone within 4 weeks prior to day 1, intended for the treatment of prostate cancer.
* Subject received treatment with herbal medications that have known hormonal antiprostate cancer activity and/or are known to decrease PSA levels within 4 weeks prior to day 1.
* Subject received prior aminoglutethimide, ketoconazole, abiraterone acetate or enzalutamide for the treatment of prostate cancer or participation in a clinical study of an investigational agent that inhibits the AR or androgen synthesis (e.g., TAK-700, ARN-509, ODM-201).
* Subject has known or suspected brain metastasis or active leptomeningeal disease.
* Subject has absolute neutrophil count < 1500/μL, platelet count < 100000/μL or hemoglobin < 10 g/dL (6.2 mmol/L).
* Subject has total bilirubin (TBL) ≥ 1.5 x the upper limit of normal (ULN) (except subjects with documented Gilbert's disease), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 x the ULN .
* Subject has creatinine > 2 mg/dL (177 μmol/L).
* Subject has albumin < 3.0 g/dL (30 g/L).
* Subject has a history of seizure or any condition that may predispose to seizure.
* Subject has history of loss of consciousness or transient ischemic attack within 12 months prior to day 1.
* Subject has clinically significant cardiovascular disease.
* Subject received bisphosphonates or denosumab within 2 weeks prior to day 1 unless administered at stable dose or to treat diagnosed osteoporosis

Exclusion Criteria for Open-Label Extension:

* Subject has taken commercially available enzalutamide (Xtandi).
* Subject's disease has progressed radiographically during the double-blind period of the study and treatment with study drug was stopped prior to study-wide unblinding. (Note: Subjects who progressed radiographically while in the double-blind portion of the study and continued treatment per protocol are allowed to participate in the open label extension.)
* After study-wide unblinding, subject has started any new investigational agent or anti-neoplastic therapy intended to treat prostate cancer
* Subject has any clinically significant disorder or condition including excessive alcohol or drug abuse, or secondary malignancy, which may interfere with study participation
* Subject has current or previously treated brain metastasis or active leptomeningeal disease
* Subject has a history of seizure or any condition that may increase the risk of seizure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (203):
- United States (34):
  - Site US10016, Homewood, Alabama
  - Site US10007, Anchorage, Alaska
  - Site US10008, Tucson, Arizona
  - Site US10034, Fountain Valley, California
  - Site US10056, La Jolla, California
  - Site US10026, Santa Rosa, California
  - Site US10035, Aurora, Colorado
  - Site US10050, Denver, Colorado
  - Site US10048, St. Petersburg, Florida
  - Site US10054, Thomasville, Georgia
  - Site US10015, Chicago, Illinois
  - Site US10043, Springfield, Illinois
  - Site US10045, Jeffersonville, Indiana
  - Site US10020, West Des Moines, Iowa
  - Site US10055, Kansas City, Kansas
  - Site US10017, Towson, Maryland
  - Site US10036, Omaha, Nebraska
  - Site US10018, Lawrenceville, New Jersey
  - Site US10025, Newburgh, New York
  - Site US10029, Syracuse, New York
  - Site US10068, Charlotte, North Carolina
  - Site US10009, Concord, North Carolina
  - Site US10014, Durham, North Carolina
  - Site US10060, Greenville, North Carolina
  - Site US10044, Middleburg Heights, Ohio
  - Site US10011, Lancaster, Pennsylvania
  - Site US10012, Myrtle Beach, South Carolina
  - Site US10059, Nashville, Tennessee
  - Site US10046, Dallas, Texas
  - Site US10004, Dallas, Texas
  - Site US10040, Virginia Beach, Virginia
  - Site US10002, Burien, Washington
  - Site US10013, Seattle, Washington
  - Site US10028, Wenatchee, Washington
- Argentina (3):
  - Site AR54002, Rosario, Santa Fe Province
  - Site AR54007, San Miguel de Tucumán, Tucumán Province
  - Site AR54010, Buenos Aires
- Australia (10):
  - Site AU61016, Camperdown, New South Wales
  - Site AU61007, St Leonards, New South Wales
  - Site AU61006, Sydney, New South Wales
  - Site AU61009, Tweed Heads, New South Wales
  - Site AU61013, Waratah, New South Wales
  - Site AU61001, Woodville South, South Australia
  - Site AU61004, Ballarat, Victoria
  - Site AU61015, Clayton, Victoria
  - Site AU61017, Parkville, Victoria
  - Site AU61008, St Albans, Victoria
- Belgium (5):
  - Site BE32001, Mons, Hainaut
  - Site BE32012, Ghent, Oost-Vlaanderen
  - Site BE32005, Kortrijk, West-Vlaanderen
  - Site BE32008, Liège
  - Site BE32007, Yvoir
- Canada (10):
  - Site CA15016, Edmonton, Alberta
  - Site CA15024, Abbotsford, British Columbia
  - Site CA15003, Kelowna, British Columbia
  - Site CA15022, Kelowna, British Columbia
  - Site CA15010, Brampton, Ontario
  - Site CA15021, Kingston, Ontario
  - Site CA15013, Oakville, Ontario
  - Site CA15020, Toronto, Ontario
  - Site CA15023, Granby, Quebec
  - Site CA15004, Montreal, Quebec
- Chile (6):
  - Site CL56002, Temuco, Región de la Araucanía
  - Site CL56005, Viña del Mar, Región de Valparaíso
  - Site CL56001, Santiago, RM
  - Site CL56007, Providencia, Santiago Metropolitan
  - Site CL56004, Reñaca, Viña Del Mar
  - Site CL56003, Santiago
- Denmark (6):
  - Site DK45005, Aarhus, Central Jutland
  - Site DK45008, Holstebro, Central Jutland
  - Site DK45002, Copenhagen, Hovestaden
  - Site DK45004, Aalborg, North Denmark
  - Site DK45003, Herlev
  - Site DK45001, Odense C
- Finland (7):
  - Site FI35802, Helsinki, Etelä-Suomen Lääni
  - Site FI35804, Pori, Länsi-Suomen Lääni
  - Site FI35803, Seinäjoki, Länsi-Suomen Lääni
  - Site FI35801, Tampere, Oulun Laani
  - Site FI35806, Jakobstad
  - Site FI35805, Oulu
  - Site FI35807, Turku
- France (12):
  - Site FR33010, Angers, Maine-et-Loire
  - Site FR33003, Créteil, Val-de-Marne
  - Site FR33006, Bordeaux
  - Site FR33014, Caen
  - Site FR33005, La Roche-sur-Yon
  - Site FR33015, Le Mans
  - Site FR33012, Lille
  - Site FR33007, Lyon
  - Site FR33011, Nîmes
  - Site FR33001, Pierre-Bénite
  - Site FR33009, Quimper
  - Site FR33013, Saint-Mandé
- Germany (5):
  - Site DE49002, Freiburg im Breisgau, Baden-Wurttemberg
  - Site DE49004, Nürtingen, Baden-Wurttemberg
  - Site DE49005, Bonn
  - Site DE49014, Hamburg
  - Site DE49013, Heidelberg
- Israel (6):
  - Site IL97201, Kfar Saba, Central District
  - Site IL97211, Ẕerifin, Central District
  - Site IL97210, Beersheba
  - Site IL97202, Haifa
  - Site IL97205, Haifa
  - Site IL97206, Jerusalem
- Italy (9):
  - Site IT39005, Meldola, Emilia-Romagna
  - Site IT39004, Cremona, Lombardy
  - Site IT39003, Milan, Lombardy
  - Site IT39012, Milan, Lombardy
  - Site IT39007, Novara, Piedmont
  - Site IT39011, Trento, Trentino-Alto Adige
  - Site IT39008, Pisa, Tuscany
  - Site IT39006, Padua, Veneto
  - Site IT39009, Candiolo
- Japan (19):
  - Site JP81003, Sakura, Chiba
  - Site JP81001, Maebashi, Gunma
  - Site JP81013, Kita-gun, Kagawa-ken
  - Site JP81007, Yokohama, Kanagawa
  - Site JP81016, Sendai, Miyagi
  - Site JP81010, Abeno-ku, Osaka
  - Site JP81011, Chuo-ku, Osaka
  - Site JP81012, Sayama, Osaka
  - Site JP81006, Bunkyo-ku, Tokyo
  - Site JP81004, Koto-ku, Tokyo
  - Site JP81005, Shinjuku-ku, Tokyo
  - Site JP81017, Ube, Yamaguchi
  - Site JP81002, Chiba
  - Site JP81014, Fukuoka
  - Site JP81015, Fukuoka
  - Site JP81008, Kyoto
  - Site JP81018, Nagasaki
  - Site JP81020, Niigata
  - Site JP81019, Yamagata
- Netherlands (8):
  - Site NL31003, Nijmegen, Gelderland
  - Site NL31007, Nijmegen, Gelderland
  - Site NL31005, Eindhoven, North Brabant
  - Site NL31010, Alkmaar, North Holland
  - Site NL31008, Amsterdam, North Holland
  - Site NL31009, Zwolle, Overijssel
  - Site NL31002, Sneek, Provincie Friesland
  - Site NL31006, Rotterdam, South Holland
- New Zealand (5):
  - Site NZ64003, Tauranga, Bay of Plenty
  - Site NZ64008, Kensington, Northland
  - Site NZ64002, Dunedin, South Island
  - Site NZ64005, Nelson, Tasman District
  - Site NZ64004, Hamilton
- Poland (6):
  - Site PL48007, Krakow, Lesser Poland Voivodeship
  - Site PL48003, Wroclaw, Lower Silesian Voivodeship
  - Site PL48011, Warsaw, Masovian Voivodeship
  - Site PL48005, Gdansk, Pomeranian Voivodeship
  - Site PL48010, Słupsk, Pomeranian Voivodeship
  - Site PL48001, Mysłowice
- Romania (7):
  - Site RO40008, Cluj-Napoca, Cluj
  - Site RO40009, Cluj-Napoca, Cluj
  - Site RO40002, Floreşti, Cluj
  - Site RO40011, Timișoara, Timiș County
  - Site RO40007, Brasov
  - Site RO40003, Bucharest
  - Site RO40006, Bucharest
- Russia (11):
  - Site RU70013, Ivanovo
  - Site RU70001, Moscow
  - Site RU70003, Moscow
  - Site RU70014, Moscow
  - Site RU70006, Omsk
  - Site RU70005, Penza
  - Site RU70007, Saint Petersburg
  - Site RU70008, Saint Petersburg
  - Site RU70009, Saint Petersburg
  - Site RU70012, Saint Petersburg
  - Site RU70016, Saint Petersburg
- Slovakia (7):
  - Site SK42110, Bratislava
  - Site SK42109, Košice
  - Site SK42102, Michalovce
  - Site SK42103, Nitra
  - Site SK42101, Poprad
  - Site SK42107, Trenčín
  - Site SK42106, Žilina
- South Korea (6):
  - Site KR82008, Seongnam-si, Gyeonggi-do
  - Site KR82007, Busan
  - Site KR82004, Incheon
  - Site KR82001, Seoul
  - Site KR82002, Seoul
  - Site KR82003, Seoul
- Spain (11):
  - Site ES34011, Salamanca, A Coruña
  - Site ES34010, Sabadell, Barcelona
  - Site ES34012, Barcelona, Catalonia
  - Site ES34014, Barcelona, Catalonia
  - Site ES34006, Pamplona, Navarre
  - Site ES34020, Oviedo, Principality of Asturias
  - Site ES34013, Valencia, Valencia
  - Site ES34001, Ávila
  - Site ES34007, Barcelona
  - Site ES34004, Madrid
  - Site ES34019, Madrid
- Sweden (5):
  - Site SE46002, Örebro, Orebro Län
  - Site SE46001, Malmo, Skåne County
  - Site SE46006, Stockholm, Södermanland County
  - Site SE46004, Sundsvall, Västernorrland County
  - Site SE46007, Gothenburg, Västra Götaland County
- Taiwan (4):
  - Site TW88601, Kaohsiung City
  - Site TW88606, Taichung
  - Site TW88605, Taipei
  - Site TW88607, Taoyuan District
- Site GB44002, Withington, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Result] Armstrong AJ, Szmulewitz RZ, Petrylak DP, Holzbeierlein J, Villers A, Azad A, Alcaraz A, Alekseev B, Iguchi T, Shore ND, Rosbrook B, Sugg J, Baron B, Chen L, Stenzl A. ARCHES: A Randomized, Phase III Study of Androgen Deprivation Therapy With Enzalutamide or Placebo in Men With Metastatic Hormone-Sensitive Prostate Cancer. J Clin Oncol. 2019 Nov 10;37(32):2974-2986. doi: 10.1200/JCO.19.00799. Epub 2019 Jul 22. PMID 31329516
- [Derived] Azad AA, Petrylak DP, Iguchi T, Shore ND, Villers A, Gomez-Veiga F, Alcaraz A, Alekseev B, Szmulewitz RZ, Holzbeierlein J, Rosbrook B, Ma J, Zohren F, El-Chaar NN, Haas GP, Stenzl A, Armstrong AJ. Enzalutamide and Prostate-Specific Antigen Levels in Metastatic Prostate Cancer: A Secondary Analysis of the ARCHES Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e258751. doi: 10.1001/jamanetworkopen.2025.8751. PMID 40332939
- [Derived] Armstrong AJ, Azad AA, Conduit C, Haas GP, Bland C, Davis ID. Enzalutamide in metastatic hormone-sensitive prostate cancer: A plain language summary of the ARCHES and ENZAMET follow-up studies. Future Oncol. 2025 Jan;21(1):15-24. doi: 10.1080/14796694.2024.2408101. Epub 2024 Oct 15. PMID 39404227
- [Derived] Armstrong AJ, Iguchi T, Azad AA, Villers A, Alekseev B, Petrylak DP, Szmulewitz RZ, Alcaraz A, Shore ND, Holzbeierlein J, Gomez-Veiga F, Rosbrook B, Zohren F, Haas GP, Gourgiotti G, El-Chaar N, Stenzl A. The Efficacy of Enzalutamide plus Androgen Deprivation Therapy in Oligometastatic Hormone-sensitive Prostate Cancer: A Post Hoc Analysis of ARCHES. Eur Urol. 2023 Aug;84(2):229-241. doi: 10.1016/j.eururo.2023.04.002. Epub 2023 May 12. PMID 37179240
- [Derived] Cella D, Ganguli A, Turnbull J, Rohay J, Morlock R. US Population Reference Values for Health-Related Quality of Life Questionnaires Based on Demographics of Patients with Prostate Cancer. Adv Ther. 2022 Aug;39(8):3696-3710. doi: 10.1007/s12325-022-02204-3. Epub 2022 Jun 22. PMID 35731340
- [Derived] Armstrong AJ, Azad AA, Iguchi T, Szmulewitz RZ, Petrylak DP, Holzbeierlein J, Villers A, Alcaraz A, Alekseev B, Shore ND, Gomez-Veiga F, Rosbrook B, Zohren F, Yamada S, Haas GP, Stenzl A. Improved Survival With Enzalutamide in Patients With Metastatic Hormone-Sensitive Prostate Cancer. J Clin Oncol. 2022 May 20;40(15):1616-1622. doi: 10.1200/JCO.22.00193. Epub 2022 Apr 14. PMID 35420921
- [Derived] Stenzl A, Dunshee C, De Giorgi U, Alekseev B, Iguchi T, Szmulewitz RZ, Flaig TW, Tombal B, Morlock R, Ivanescu C, Ramaswamy K, Saad F, Armstrong AJ. Effect of Enzalutamide plus Androgen Deprivation Therapy on Health-related Quality of Life in Patients with Metastatic Hormone-sensitive Prostate Cancer: An Analysis of the ARCHES Randomised, Placebo-controlled, Phase 3 Study. Eur Urol. 2020 Oct;78(4):603-614. doi: 10.1016/j.eururo.2020.03.019. Epub 2020 Apr 23. PMID 32336645
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/9785-CL-0335
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14403&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with metastatic hormone sensitive prostate cancer (mHSPC) were enrolled in 204 study sites worldwide.
Pre-assignment Details: The randomization was stratified by volume of disease (low vs high) and prior docetaxel therapy for prostate cancer (no prior docetaxel, 1 to 5 cycles, 6 cycles).
Groups:
- Enzalutamide + Androgen Deprivation Therapy (ADT): Participants received 160 mg of enzalutamide orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. Eligible participants who received enzalutamide during double-blind treatment period and provided informed consent to take part in open-label period continued to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or luteinizing hormone-releasing hormone (LHRH) agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
- Placebo + Androgen Deprivation Therapy (ADT): Participants received enzalutamide matching placebo orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. Eligible participants who received enzalutamide matching placebo during double-blind treatment period and provided informed consent to take part in open-label period switched to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
Period: Double Blind Period (up to 35 Months)
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Started | 574 | 576
Treated | 572 | 574
Completed | 0 | 0
Not Completed | 574 | 576
Not completed — Death | 117 | 197
Not completed — Lost to Follow-up | 12 | 15
Not completed — Progressive disease | 3 | 6
Not completed — Withdrawal by Subject | 41 | 71
Not completed — Miscellaneous | 30 | 99
Not completed — Continued in OLE | 370 | 182
Not completed — Discontinued by Sponsor | 1 | 4
Not completed — Randomized, Not Treated | 0 | 2
Period: Open-Label Extension (Approx. 66 Months)
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Started | 370 (Eligible participants who provided consent took part in open-label period) | 182 (Eligible participants who provided consent took part in open-label period)
Completed | 0 | 0
Not Completed | 370 | 182
Not completed — Death | 73 | 26
Not completed — Lost to Follow-up | 8 | 3
Not completed — Progressive disease | 22 | 10
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Miscellaneous | 241 | 125
Not completed — Discontinued by Sponsor | 10 | 5

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Enzalutamide + Androgen Deprivation Therapy (ADT): Participants received 160 mg of enzalutamide orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. Eligible participants who received enzalutamide during double-blind treatment period and provided informed consent to take part in open-label period continued to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock.
- Total: Total of all reporting groups
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT) | Total
Number analyzed (Participants) | 574 | 576 | 1150
Age, Continuous [Mean (Standard Deviation); unit: year] | 69.5 (8.0) | 69.5 (8.4) | 69.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 574 | 576 | 1150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 37 | 83
  Not Hispanic or Latino | 504 | 514 | 1018
  Unknown or Not Reported | 24 | 25 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 75 | 80 | 155
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 466 | 460 | 926
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 28 | 53
Volume of Disease [Count of Participants; unit: Participants] — High volume of disease was defined as metastases involving the viscera or, in the absence of visceral lesions, 4 or more bone lesions, at least 1 of which was in a bony structure beyond the vertebral column and pelvic bone. Low volume was anything that wasn't considered high volume by definition provided. Population: Intent-to-Treat (ITT)
  Participants
    Low | 220 | 203 | 423
    High | 354 | 373 | 727
Prior Docetaxel Therapy Use [Count of Participants; unit: Participants] — Population: ITT
  Participants
    None | 471 | 474 | 945
    1 to 5 cycles | 14 | 11 | 25
    6 cycles | 89 | 91 | 180

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival (rPFS) Based on Independent Central Review (ICR) of Bone Scan According to Prostate Cancer Clinical Trials Working Group 2 (PCWG2) Criteria
Description: rPFS was calculated as the time from the date of randomization to the first objective evidence of radiographic progression disease (rPD) at any time or death up to 24 weeks after study drug discontinuation without documented radiographic progression, whichever occurred first. rPD was defined as progressive disease by Response Evaluation Criteria in Solid Tumors version 1.1 for soft tissue disease or by appearance of 2 or more new lesions on bone scan compared to baseline or week 13 according to PCWG2 criteria, as assessed by ICR or death. In participants with no rPFS event, rPFS was censored on the date of last evaluable radiographic assessment prior to the data analysis cutoff date. In participants with no baseline radiographic assessment, participants with no postbaseline radiographic assessments and participants with all postbaseline radiographic assessments documented as "not evaluable (NE)," rPFS was censored on the date of randomization.
Time Frame: From the date of randomization to the first objective evidence of rPD at any time or death (maximum duration was 26.6 months)
Population: ITT population is defined as all participants who were randomized in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | 19.4 [16.59 to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); rPFS Treatment Comparison; Test type: Superiority; p < 0.0001, Log Rank — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox hazard ratio = 0.39, 95% CI 2-sided [0.30 to 0.50] — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period

2. Primary Outcome: rPFS Based on ICR of Bone Scan According to Protocol Assessment Criteria
Description: rPFS was calculated as the time from the date of randomization to the first objective evidence of radiographic progression disease (rPD) at any time or death up to 24 weeks after study drug discontinuation without documented radiographic progression, whichever occurred first. rPD was defined as progressive disease by Response Evaluation Criteria in Solid Tumors version 1.1 for soft tissue disease or by appearance of 2 or more new lesions on bone scan compared to baseline for week 13 or the best response on treatment for week 25 or later assessments, as assessed by ICR or death. In participants with no rPFS event, rPFS was censored on the date of last evaluable radiographic assessment prior to the data analysis cutoff date. In participants with no baseline radiographic assessment, participants with no postbaseline radiographic assessments and participants with all postbaseline radiographic assessments documented as "not evaluable (NE)," rPFS was censored on the date of randomization.
Time Frame: as for outcome 1
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | 19.0 [16.59 to 22.24]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); rPFS Treatment Comparision; Test type: Superiority; p < 0.0001, Log Rank; Cox proportional hazards model = 0.39, 95% CI 2-sided [0.30 to 0.50]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. In participants still alive at the date of the analysis cutoff point, OS was censored on the last date the participant was known to be alive. OS was analyzed using Kaplan-Meier estimates.
Time Frame: From randomization to death due to any cause (maximum duration was 58.6 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | NA [49.74 to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Test type: Superiority; p < 0.0001, Log Rank; P-value from stratified log-rank test; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.53 to 0.81] — Significance level is 0.04. Hazard ratio and 95 % CI are estimated by cox proportional hazards model

4. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression
Description: Time to PSA progression was calculated as the time from the date of randomization to the first observation of PSA progression. A PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir, which was confirmed by a second consecutive value at least 3 weeks later. In participants with no PSA progression, time to PSA progression was censored on the date of the last PSA sample taken (or last value prior to 2 or more consecutive missed PSA assessments).
Time Frame: From the date of randomization to the first observation of PSA progression (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | NA [16.59 to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to PSA Progression Treatment Comparison; Test type: Superiority; p < 0.0001, Log Rank — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox hazard ratio = 0.19, 95% CI 2-sided [0.13 to 0.26] — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period

5. Secondary Outcome: Time to Start of New Antineoplastic Therapy
Description: In participants with a new antineoplastic therapy initiated for prostate cancer after randomization, time to start of a new antineoplastic therapy was defined as the time interval from randomization to the date of the first dose administration of the first antineoplastic therapy. In participants with no new antineoplastic therapy initiated for prostate cancer after randomization, time to start of new antineoplastic therapy was censored on the last visit date or the date of randomization, whichever occurred last. Time to start of new antineoplastic therapy was analyzed using Kaplan-Meier estimates.
Time Frame: From randomization to the date of the first dose administration of the first antineoplastic therapy (maximum duration was 58.6 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | 40.5 [26.25 to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Test type: Superiority; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.31 to 0.48] — Hazard ratio and 95 % CI are estimated by cox proportional hazards model

6. Secondary Outcome: PSA Undetectable Rate
Description: The PSA undetectable rate was defined as the percentage of participants with undetectable (< 0.2 ng/mL) PSA values at any time during study treatment, of those participants with detectable (≥ 0.2 ng/mL) PSA values at baseline.
Time Frame: From baseline to detectable PSA values (maximum duration was 26.6 months)
Population: ITT with detectable PSA at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 511 | 506
percentage of participants | 68.1 [63.9 to 72.1] | 17.6 [14.4 to 21.2]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); PSA Undetectable Rate Treatment Comparison; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Difference in rate = 50.5, 95% CI 2-sided [45.3 to 55.7]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was calculated as the percentage of participants who achieved a completed response (CR) or a partial response (PR) (unconfirmed responses) in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by ICR.
Time Frame: From date of randomization up to 26.6 months
Population: ITT participants with measurable disease at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 177 | 182
percentage of participants | 83.1 [76.7 to 88.3] | 63.7 [56.3 to 70.7]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); ORR Treatment Comparison; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Difference in rate = 19.3, 95% CI 2-sided [10.4 to 28.2]

8. Secondary Outcome: Time to Deterioration in Urinary Symptoms
Description: In participants with deterioration, the time to deterioration was calculated as the time interval between randomization and the first deterioration in urinary symptoms at any postbaseline visit. A deterioration in urinary symptoms was defined as an increase in the Quality of Life Prostate-specific Questionnaire (QLQ-PR25) modified urinary symptoms. Subscale score by ≥ 50% of the standard deviation observed in the QLQ-PR25 modified urinary symptoms subscale score at baseline. Modified urinary symptoms subscale score consisted of 3-items (Q31 - Q33) from the QLQ-PR25, each scored from 1 (not at all) to 4 (very much). The total modified urinary symptoms subscale score ranges from 0-100, with higher scores represents a higher level of symptomatology/problems. In participants without deterioration in urinary symptoms, the time to deterioration in urinary symptoms was censored on the date the last urinary symptoms QLQ-PR25 score was calculable.
Time Frame: From date of randomization to the first deterioration in urinary symptoms at any postbaseline visit (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [19.35 to NA] — Not reached. Data was not reached due to low number of events. | 16.8 [14.06 to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to Deterioration of Urinary Symptoms Treatment Comparison; Test type: Superiority; p = 0.2162, Log Rank — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox hazard ratio = 0.88, 95% CI 2-sided [0.72 to 1.08] — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period

9. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: Time to first SSE was calculated as the time from randomization to the occurrence of the first SSE. An SSE was defined as radiation to bone, surgery to bone, clinically apparent pathological bone fracture, or spinal cord compression. In participants with no SSE, time to SSE was censored on the last visit date or the date of randomization, whichever occurred last.
Time Frame: From randomization to the occurrence of the first SSE (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | NA [NA to NA] — Not reached. Data was not reached due to low number of events.
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to SSE Treatment Comparison; Test type: Superiority; p = 0.0026, Log Rank; Cox hazard ratio = 0.52, 95% CI 2-sided [0.33 to 0.80]

10. Secondary Outcome: Time to Castration Resistance
Description: Time to castration resistance was calculated as the time from randomization to the first castration-resistant event. A castration resistance event was defined as any of the following in the presence of castrate levels of testosterone (< 50 ng/dL): radiographic disease progression, PSA progression or SSE, whichever occurred first. In participants with no documented castration resistance event, the time to castration resistance was censored on the latest date from: the date of last radiologic assessment, the last PSA sample taken prior to the start of any new prostate cancer therapy and prior to 2 or more consecutive missed PSA assessments (if applicable), and the last visit date performed.
Time Frame: From randomization to the first castration-resistant event (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | NA [NA to NA] — Not reached. Data was not reached due to low number of events. | 13.9 [11.40 to 17.18]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to Castration Resistance Treatment Comparison; Test type: Superiority; p < 0.0001, Log Rank; Cox hazard ratio = 0.28, 95% CI 2-sided [0.22 to 0.36]

11. Secondary Outcome: Time to Deterioration of Quality of Life (QoL) in Functional Assessment of Cancer Therapy-Prostate (FACT-P)
Description: Time to deterioration of QoL was calculated as the time interval from the date of randomization to the first date a decline from baseline of 10 points or more in the FACT-P total score was recorded. The FACT-P consists of 27 core items that assess participant function in 4 domains and 12 prostate cancer-related items grouped into 5 subscales as follows: physical wellbeing, social/family wellbeing, emotional wellbeing, functional wellbeing and prostate cancer subscale. Each item is rated on a 0 to 4 Likert-type scale. The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0 to 156), where high score represent better quality of life. In participants without FACT-P progression, the time to deterioration of QoL was censored on the date of the last FACT-P total score was calculable.
Time Frame: From the date of randomization to the first date a decline from baseline of 10 points or more in the FACT-P total score (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | 11.3 [11.04 to 13.83] | 11.1 [8.48 to 13.83]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to Deterioration of QoL in FACT-P Treatment Comparison; Test type: Superiority; p = 0.6548, Log Rank; Cox hazard ratio = 0.96, 95% CI 2-sided [0.81 to 1.14]

12. Secondary Outcome: Time to Pain Progression Based on Brief Pain Inventory-Short Form (BPI-SF)
Description: Time to pain progression was defined as time from randomization to the first pain progression event. Pain progression was defined as an increase of ≥ 30% from baseline in the average BPI-SF pain severity score. BPI-SF contains 9 questions with rating scales from 0 (no pain/no interference) to 10 (worst pain/interferes completely). Total score was calculated as the average of each question. Higher scores represent a higher level of pain or interference. In participants with no pain progression event, time to pain progression was censored on the last visit date where BPI-SF was collected.
Time Frame: From randomization to the first pain progression event (maximum duration was 26.6 months)
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 574 | 576
months | 8.3 [8.25 to 10.91] | 8.3 [5.65 to 8.38]
Statistical Analysis 1: Comparison: Enzalutamide + Androgen Deprivation Therapy (ADT) vs Placebo + Androgen Deprivation Therapy (ADT); Time to Pain Progression Based on BPI-SF Treatment Comparison; Test type: Superiority; p = 0.2715, Log Rank; Cox hazard ratio = 0.92, 95% CI 2-sided [0.78 to 1.07]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization up to end of study duration (approximately 7 years) AEs: From first dose up to 30 days after last dose of study drug (maximum duration of treatment 7 years)
Description: All-cause mortality: The at risk population included all randomized participants
  AEs: The at risk population included the Safety Analysis Set (SAF) consisting of all randomized participants who received at least one dose of study drug.
Groups:
- Placebo + ADT: Participants received enzalutamide matching placebo orally once daily during double-blind treatment period until radiographic progression was documented or until the participants started an investigational agent or new therapy for treatment of prostate cancer or until any other discontinuation criterion was met. This arm represents only double blind period.
- Placebo Cross-over Enzalutamide: Eligible participants who received enzalutamide matching placebo during double-blind treatment period and provided informed consent to take part in open-label period switched to receive 160 mg enzalutamide orally once daily in open-label period until disease progression, unacceptable toxicity or any other discontinuation criteria were met. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment as per standard of care and provided by the site's pharmacy stock. This arm represents only the open-label extension period.
Arm/Group | Enzalutamide + Androgen Deprivation Therapy (ADT) | Placebo + ADT | Placebo Cross-over Enzalutamide
All-Cause Mortality (participants affected / at risk) | 190/574 | 197/576 | 27/182
Serious Adverse Events (participants affected / at risk) | 244/572 | 128/574 | 81/182
Other Adverse Events (participants affected / at risk) | 463/572 | 401/574 | 133/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Androgen Deprivation Therapy (ADT) (N=572) | Placebo + ADT (N=574) | Placebo Cross-over Enzalutamide (N=182)
Anaemia (Blood and lymphatic system disorders) | 7 (11) | 2 (4) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (6) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 4 (8) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (13) | 7 (10) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 6 (8) | 1 (1) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 5 (7)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (4) | 1 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (5) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 2 (3) | 2 (3)
Implant site dehiscence (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (2)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 3 (5)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 7 (12) | 0 (0) | 2 (3)
COVID-19 pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Genital abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 9 (13) | 5 (6) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 3 (3) | 2 (3)
Septic shock (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 12 (12) | 4 (4) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 2 (3)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 2 (2)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 3 (3)
Stenosis of vesicourethral anastomosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrong dose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Antineutrophil cytoplasmic antibody increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Blood testosterone increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (5) | 2 (4)
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (5) | 1 (2)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (4)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (2)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (10) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (14) | 3 (4) | 4 (6)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (4) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (6) | 1 (1) | 3 (3)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 3 (3) | 7 (7) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 2 (3) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (11) | 3 (3) | 1 (3)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (13) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 3 (4) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 9 (9) | 4 (4) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 2 (2)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3) | 5 (6)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2)
Bone lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Aortic dissection rupture (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 3 (7)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (3) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac pseudoaneurysm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Flail chest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of personal independence in daily activities (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide + Androgen Deprivation Therapy (ADT) (N=572) | Placebo + ADT (N=574) | Placebo Cross-over Enzalutamide (N=182)
Anaemia (Blood and lymphatic system disorders) | 51 (86) | 28 (39) | 5 (6)
Constipation (Gastrointestinal disorders) | 61 (72) | 34 (34) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 56 (72) | 34 (35) | 9 (10)
Nausea (Gastrointestinal disorders) | 54 (65) | 34 (35) | 14 (19)
Asthenia (General disorders) | 52 (79) | 29 (36) | 6 (7)
Fatigue (General disorders) | 147 (197) | 92 (103) | 43 (54)
Oedema peripheral (General disorders) | 51 (66) | 40 (48) | 8 (9)
Nasopharyngitis (Infections and infestations) | 55 (74) | 33 (39) | 14 (22)
Fall (Injury, poisoning and procedural complications) | 63 (96) | 16 (16) | 19 (30)
Weight increased (Investigations) | 46 (89) | 45 (51) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 43 (46) | 18 (20) | 15 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 147 (214) | 79 (99) | 19 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 89 (128) | 66 (69) | 29 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 35 (45) | 30 (33) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 (48) | 27 (28) | 11 (12)
Dizziness (Nervous system disorders) | 47 (50) | 22 (24) | 9 (9)
Headache (Nervous system disorders) | 52 (62) | 22 (27) | 8 (9)
Insomnia (Psychiatric disorders) | 32 (36) | 21 (22) | 6 (6)
Gynaecomastia (Reproductive system and breast disorders) | 34 (39) | 8 (8) | 4 (4)
Hot flush (Vascular disorders) | 172 (199) | 131 (137) | 16 (18)
Hypertension (Vascular disorders) | 88 (107) | 36 (38) | 19 (22)
COVID-19 (Infections and infestations) | 29 (30) | 0 (0) | 18 (20)
Rib fracture (Injury, poisoning and procedural complications) | 38 (47) | 6 (8) | 12 (18)
Weight decreased (Investigations) | 30 (39) | 16 (17) | 14 (15)
Haematuria (Renal and urinary disorders) | 34 (45) | 13 (15) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02677896/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT02677896/SAP_003.pdf